CLINICAL TRIAL: NCT05681767
Title: Motivational Multicomponent Lifestyle Interventions as a Supportive Treatment for Depression in Primary Health Care
Acronym: DEPKuopio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); City of Kuopio (Other Government); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH500SH07
Record Dates: First submitted 2022-12-09; First posted 2023-01-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a 2-arm, randomized controlled clinical trial, in which participants are randomized to the study arms at an individual level. After the baseline data is collected, the study nurse (nurse 1), who conducts the baseline data collection, uses opaque capsules to randomize patients to the study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Motivational multicomponent lifestyle intervention + treatment as usual
  Interventions: Behavioral: Motivational multicomponent lifestyle intervention + Treatment as usual
- Control group (Other): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Motivational multicomponent lifestyle intervention + Treatment as usual — Study intervention and treatment as usual
  The study intervention is a multicomponent lifestyle intervention that targets exercise, diet, and stress management, and is conducted by motivational interviewing. The study nurse provides the study intervention. The intervention is conducted by motivational interviewing and includes the key elements of lifestyle interventions identified as effective (assessment of behavior at the baseline, giving information and advising, individualized goal setting, setting an action plan, monitoring a behavioral change, and giving feedback).
  The intervention consists of individual appointments (2 x 45-60 min) and a telephone session ( 2 x 15 min) for three months. The participants receive a short educational guide (A4) on the lifestyle behavior recommendations.
  Arms: Intervention group
Other: Treatment as usual — Treatment as usual
  Arms: Control group

SUMMARY:
The investigators aim to examine whether a motivational multicomponent lifestyle intervention as a supportive treatment for depression has a beneficial effect on recovery from depression in a primary health care setting.

DETAILED DESCRIPTION:
Depression causes a significant global burden of disease. Among depressed individuals, poor lifestyles, such as physical inactivity, unhealthy diet, and smoking, are common and play a role in the development and maintenance of depression. Robust research evidence recommends applying one-component lifestyle interventions that focus on factors such as a healthy diet or exercise, as a supportive treatment for depression. Currently, however, there is increasing interest in identifying the most effective multicomponent lifestyle intervention that targets more than one unhealthy lifestyle simultaneously in order to reduce depressive symptoms.

The study aims to examine whether a motivational multicomponent lifestyle intervention as a supportive treatment for depression has a beneficial effect on recovery from depression in a primary health care setting. The specific study questions are as follows:

1. What is the effect of the intervention on depressive symptoms at 3- and 12-month follow-ups?
2. What is the effect of the intervention on mental well-being at 3- and 12-month follow-ups?
3. What kind of physical health do depressed patients in primary health care have? What kinds of effects does the intervention have on common physical health risk factors at 12- and 24- month follow-ups?
4. What is the effect of the intervention on health-related quality of life?
5. What is the cost-effectiveness of the intervention?

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years
* depression (ICD-10, F32-F33)
* Beck Depression Inventory (BDI-1A) ≥ 10 points
* the initiation of treatment in a primary health care center

Exclusion Criteria:

* bipolar disorder
* psychosis
* substance abuse
* pregnancy or lactation
* a long-term rehabilitative psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory (BDI) scores | Change from baseline at 3, 12 and 24 months
  Depressive symptoms
Change in the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) scores | Change from baseline at 3, 12 and 24 months
  Mental Wellbeing
Change in 15D scores | Change from baseline at 3, 12 and 24 months
  Health-Related Quality of Life

SECONDARY OUTCOMES:
Change in Perceived Stress Scale (PSS-10) scores | Change from baseline at 3, 12 and 24 months
  Stress
Change in Insomnia Severity Index (ISI) scores | Change from baseline at 3, 12 and 24 months
  Insomnia
Change in Numeric Rating Scale for pain | Change from baseline at 3, 12 and 24 months
  Pain
Change in Overall Anxiety Severity and Impairment Scale (OASIS) scores | Change from baseline at 3, 12 and 24 months
  Anxiety
Change in Blood lipid levels | Change from baseline at 12 and 24 months
  P-Kol, P-KOL-LDL, P-KOL-HDL, P-Trigly
Change in weight/body mass index (BMI) | Change from baseline at 3, 12 and 24 months
  Change in measured weight/BMI
Change in waist circumference | Change from baseline at 3, 12 and 24 months
  Waist (centimeters)
Change in Blood pressure (diastolic and systolic) | Change from baseline at 3, 12, and 24 months
  Blood pressure (diastolic and systolic)
Change in Blood glucose levels | Change from baseline at 12 and 24 months
  P-Glucose and glycated haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Mäntyselkä, Principal Investigator — University of Eastern Finland
Locations (1):
- Kuopio Health Center, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No